CLINICAL TRIAL: NCT04274270
Title: Safety and Efficacy of Sequential Stereotactic Radiotherapy With S1 Combined With Endostar in the Treatment of Stage IV Lung Squamous Cell Carcinoma: Prospective, Multicenter, Exploratory Study
Brief Title: SBRT With S1 Combined With Endostar in the Treatment of Lung Cancer
Acronym: SBRTLCES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Mianyang Central Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Peking University Cancer Hospital & Institute (Other); Peking University International Hospital (Other); China-Japan Friendship Hospital (Other); Beijing 302 Hospital (Other); Second Hospital of Shanxi Medical University (Other); Qingdao Hiser Medical Group (Other); Guangxi Ruikang Hospital (Other); Panjin Liaohe Oilfield Gem Flower Hospital (Other); Tang-Du Hospital (Other); Third Affiliated Hospital of Guizhou Medical University (Unknown); Liuzhou Workers' Hospital (Other Government); The Affiliated Hospital of Xuzhou Medical University (Other); Dalian municipal central hospital affiliated of dalian medical university (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-CKES-LUNG
Record Dates: First submitted 2020-02-10; First posted 2020-02-18 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-02

CONDITIONS: Radiotherapy Side Effect
Keywords: lung cancer, SBRT, s1,endostar
MeSH Terms: conditions — Radiation Injuries; Lung Neoplasms | interventions — endostar protein; S 1 (combination)

STUDY DESIGN:
Intervention Model Description: Radiotherapy was performed with a cyberknife or accelerator stereotactic radiotherapy, which lasted 3-10 days.After the end of radiotherapy,S1 60mg, BID, day 1-28, as taken orally, and repeated every 6 weeks, with concurrent Endostar therapy: 210mg was used by intravenous infusion for 7 consecutive days during each cycle of chemotherapy, and 30mg was used every 24 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Radiotherapy was performed with a cyberknife or accelerator stereotactic radiotherapy, which lasted 3-10 days.After the end of radiotherapy,S1 60mg, BID, day 1-28, as taken orally, and repeated every 6 weeks, with concurrent Endostar therapy: 210mg was used by intravenous infusion for 7 consecutive days during each cycle of chemotherapy, and 30mg was used every 24 hours.
  Interventions: Drug: Endostar

INTERVENTIONS:
Drug: Endostar — Radiotherapy was performed with a cyberknife or accelerator stereotactic radiotherapy, which lasted 3-10 days.After the end of radiotherapy,S1 60mg, BID, day 1-28, as taken orally, and repeated every 6 weeks, with concurrent Endostar therapy: 210mg was used by intravenous infusion for 7 consecutive days during each cycle of chemotherapy, and 30mg was used every 24 hours.
  Other Names: S1

SUMMARY:
Human recombinant endostatin preclinical studies have shown that the drug can inhibit endothelial cell proliferation, angiogenesis and tumor growth, still can directly induce lung cancer cell apoptosis, multiple clinical studies in human recombinant endostatin combined with chemotherapy treatment showed good antitumor efficacy and good safety.S1 is an oral fluorouracil derivative and an improved preparation of the antitumor drug tegafur.Multiple clinical studies have reported that S1 alone or S1 combined with chemotherapy is effective in Non small cell lung cancer(NSCLC).Unfortunately, none of the prospective clinical studies to date have systematically validated the safety and efficacy of antiangiogenic drugs combined with chemotherapy in patients with advanced pulmonary SCC.The investigators expect that endu combined with S1 will increase the efficacy of advanced lung squamous cell carcinoma.The purpose of this study was to evaluate the objective remission rate and safety of entu combined with oral S1 in the treatment of advanced lung squamous cell carcinoma.

DETAILED DESCRIPTION:
In this study, the investigatorse enrolled patients with advanced lung squamous cell carcinoma to explore the safety and efficacy of sequential local radiotherapy combined with endodontic therapy.Plan to enroll 60 cases.For those who meet the inclusion criteria, medical history collection, physical examination, hematological examination and general imaging examination shall be completed before inclusion.Radiotherapy was performed with a cyberknife or accelerator stereotactic radiotherapy, which lasted 3-10 days.After the end of radiotherapy,S1 60mg, BID, day 1-28, as taken orally, and repeated every 6 weeks, with concurrent Endostar therapy: 210mg was used by intravenous infusion for 7 consecutive days during each cycle of chemotherapy, and 30mg was used every 24 hours.Treatment-related toxicity, treatment response and survival were followed up during treatment.Drug treatment until the tumor progresses, or there is an intolerable treatment-related toxicity, or no tolerance to further treatment.The treatment lasts for up to 3 years with good toxicity tolerance.During the treatment, the dose of teggio and endu is not adjusted. If serious adverse reactions occur, the drug should be treated actively and delayed.If the investigator determines that the treatment-related toxicity cannot be tolerated, the treatment is discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Lung squamous cell carcinoma was confirmed by histopathology or cytopathology;
2. Meet AJCC(8th edition, 2018) lung cancer stage IV standard;
3. Lesions requiring SBRT;
4. Measurable lesions must have at least one evaluable lesion judged according to RECIST 1.1 standard, i.e., the longest diameter is at least 20mm);
5. Age >=18 years old;
6. KPS > = 70;
7. Life expectancy of at least 3 months;
8. Hematology, liver and kidney function and cardiopulmonary function can tolerate radiotherapy and chemotherapy.

Exclusion Criteria:

1. Lung adenocarcinoma or small cell lung cancer;
2. Previous immunotherapy;
3. Patients at risk of bleeding;
4. Patients with any other malignant tumor before or now
5. Patients diagnosed with esophagotracheal fistula,uncontrolled pleural effusion,pericardial effusion requiring repeated drainage,unhealed wounds,active gastric ulcers or fractures
6. Patients suffering from poorly controlled heart disease or clinical symptoms, such as NYHA grade II or above cardiac dysfunction;unstable angina pectoris;Myocardial infarction occurred within 1 year;supraventricular or ventricular arrhythmia needs treatment or intervention;
7. Patients with known central nervous system metastases.
8. Patients with clinically suspected central nervous system metastasis must undergo enhanced CT or MRI within 28 days prior to randomization to exclude central nervous system metastasis.
9. Pregnant or breastfeeding women;Women and men who are likely to become pregnant but do not want to use appropriate contraception;
10. Other circumstances in which the investigator decides not to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
OS | 3 years
  Overall survival
PFS | the time interval of disease progression since the date of diagnosis
  Progression-free survival

SECONDARY OUTCOMES:
LCR | 2 years
  Local control rate criteria for short-term efficacy.
Adverse reactions | 2 years
  adverse events and laboratory tests were graded according to NCI CTC AE 5.0
Qol | 2 years
  Quality of life

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The fifth medical center of PLA general hospital, Beijing, Beijing Municipality
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Guangxi ruikang hospital, Nanning, Guangxi
  - Third Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Dalian municipal central hospital affiliated of dalian medical university, Dalian, Liaoning
  - GEM flower hospital of Liaohe oil field Tang-Du Hospital, Panjin, Liaoning
  - Hiser Medical Center of Qingdao, Qingdao, Shandong
  - Second hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tangdu hospital, Xian, Shanxi
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Beijing Cancer Hospital, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking University International Hospital, Beijing

REFERENCES:
- [Background] Heist RS, Mino-Kenudson M, Sequist LV, Tammireddy S, Morrissey L, Christiani DC, Engelman JA, Iafrate AJ. FGFR1 amplification in squamous cell carcinoma of the lung. J Thorac Oncol. 2012 Dec;7(12):1775-1780. doi: 10.1097/JTO.0b013e31826aed28. PMID 23154548
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Crino L, Weder W, van Meerbeeck J, Felip E; ESMO Guidelines Working Group. Early stage and locally advanced (non-metastatic) non-small-cell lung cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2010 May;21 Suppl 5:v103-15. doi: 10.1093/annonc/mdq207. No abstract available. PMID 20555058
- [Background] Felip E, Stahel RA, Pavlidis N; ESMO Guidelines Task Force. ESMO Minimum Clinical Recommendations for diagnosis, treatment and follow-up of non-small-cell lung cancer (NSCLC). Ann Oncol. 2005;16 Suppl 1:i28-9. doi: 10.1093/annonc/mdi821. No abstract available. PMID 15888743
- [Background] William WN Jr, Lin HY, Lee JJ, Lippman SM, Roth JA, Kim ES. Revisiting stage IIIB and IV non-small cell lung cancer: analysis of the surveillance, epidemiology, and end results data. Chest. 2009 Sep;136(3):701-709. doi: 10.1378/chest.08-2968. Epub 2009 Mar 24. PMID 19318668
- [Background] D'Angelo SP, Pietanza MC, Johnson ML, Riely GJ, Miller VA, Sima CS, Zakowski MF, Rusch VW, Ladanyi M, Kris MG. Incidence of EGFR exon 19 deletions and L858R in tumor specimens from men and cigarette smokers with lung adenocarcinomas. J Clin Oncol. 2011 May 20;29(15):2066-70. doi: 10.1200/JCO.2010.32.6181. Epub 2011 Apr 11. PMID 21482987
- [Background] Socinski MA, Evans T, Gettinger S, Hensing TA, VanDam Sequist L, Ireland B, Stinchcombe TE. Treatment of stage IV non-small cell lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e341S-e368S. doi: 10.1378/chest.12-2361. PMID 23649446
- [Background] Johnson DH, Fehrenbacher L, Novotny WF, Herbst RS, Nemunaitis JJ, Jablons DM, Langer CJ, DeVore RF 3rd, Gaudreault J, Damico LA, Holmgren E, Kabbinavar F. Randomized phase II trial comparing bevacizumab plus carboplatin and paclitaxel with carboplatin and paclitaxel alone in previously untreated locally advanced or metastatic non-small-cell lung cancer. J Clin Oncol. 2004 Jun 1;22(11):2184-91. doi: 10.1200/JCO.2004.11.022. PMID 15169807
- [Background] Scagliotti G, Novello S, von Pawel J, Reck M, Pereira JR, Thomas M, Abrao Miziara JE, Balint B, De Marinis F, Keller A, Aren O, Csollak M, Albert I, Barrios CH, Grossi F, Krzakowski M, Cupit L, Cihon F, Dimatteo S, Hanna N. Phase III study of carboplatin and paclitaxel alone or with sorafenib in advanced non-small-cell lung cancer. J Clin Oncol. 2010 Apr 10;28(11):1835-42. doi: 10.1200/JCO.2009.26.1321. Epub 2010 Mar 8. PMID 20212250
- [Background] Garon EB, Ciuleanu TE, Arrieta O, Prabhash K, Syrigos KN, Goksel T, Park K, Gorbunova V, Kowalyszyn RD, Pikiel J, Czyzewicz G, Orlov SV, Lewanski CR, Thomas M, Bidoli P, Dakhil S, Gans S, Kim JH, Grigorescu A, Karaseva N, Reck M, Cappuzzo F, Alexandris E, Sashegyi A, Yurasov S, Perol M. Ramucirumab plus docetaxel versus placebo plus docetaxel for second-line treatment of stage IV non-small-cell lung cancer after disease progression on platinum-based therapy (REVEL): a multicentre, double-blind, randomised phase 3 trial. Lancet. 2014 Aug 23;384(9944):665-73. doi: 10.1016/S0140-6736(14)60845-X. Epub 2014 Jun 2. PMID 24933332
- [Background] Meng MB, Jiang XD, Deng L, Na FF, He JZ, Xue JX, Guo WH, Wen QL, Lan J, Mo XM, Lang JY, Lu Y. Enhanced radioresponse with a novel recombinant human endostatin protein via tumor vasculature remodeling: experimental and clinical evidence. Radiother Oncol. 2013 Jan;106(1):130-7. doi: 10.1016/j.radonc.2012.10.022. Epub 2013 Jan 23. PMID 23351845
- [Background] Masuda T, Watanabe M, Fujitaka K, Hamai K, Ishikawa N, Doi M, Kitaguchi S, Yamaguchi K, Sakamoto S, Horimasu Y, Miyamoto S, Nakashima T, Senoo T, Iwamoto H, Hamada H, Hattori N. Alternate-day administration of S-1 for elderly patients with advanced non-small-cell lung carcinoma: A prospective feasibility study. Mol Clin Oncol. 2018 Nov;9(5):539-544. doi: 10.3892/mco.2018.1705. Epub 2018 Aug 24. PMID 30345049
- [Background] Iwamoto Y, Mitsudomi T, Sakai K, Yamanaka T, Yoshioka H, Takahama M, Yoshimura M, Yoshino I, Takeda M, Sugawara S, Kawaguchi T, Takahashi T, Ohta M, Ichinose Y, Atagi S, Okada M, Saka H, Nakagawa K, Nakanishi Y, Nishio K. Randomized Phase II Study of Adjuvant Chemotherapy with Long-term S-1 versus Cisplatin+S-1 in Completely Resected Stage II-IIIA Non-Small Cell Lung Cancer. Clin Cancer Res. 2015 Dec 1;21(23):5245-52. doi: 10.1158/1078-0432.CCR-14-3160. Epub 2015 Aug 7. PMID 26253869
- [Background] Ohe Y, Ohashi Y, Kubota K, Tamura T, Nakagawa K, Negoro S, Nishiwaki Y, Saijo N, Ariyoshi Y, Fukuoka M. Randomized phase III study of cisplatin plus irinotecan versus carboplatin plus paclitaxel, cisplatin plus gemcitabine, and cisplatin plus vinorelbine for advanced non-small-cell lung cancer: Four-Arm Cooperative Study in Japan. Ann Oncol. 2007 Feb;18(2):317-23. doi: 10.1093/annonc/mdl377. Epub 2006 Nov 1. PMID 17079694
- [Background] Yamashita Y, Kataoka K, Ishida T, Matsuura M, Seno N, Mukaida H, Miyahara E, Miyata Y, Okita R, Shimizu K, Watari M, Okumichi T, Okada M. A feasibility study of postoperative adjuvant therapy of carboplatin and weekly paclitaxel for completely resected non-small cell lung cancer. J Thorac Oncol. 2008 Jun;3(6):612-6. doi: 10.1097/JTO.0b013e318174e05e. PMID 18520800
- [Background] Sugaya M, Uramoto H, Uchiyama A, Nagashima A, Nakanishi R, Sakata H, Nakanishi K, Hanagiri T, Yasumoto K. Phase II trial of adjuvant chemotherapy with bi-weekly carboplatin plus paclitaxel in patients with completely resected non-small cell lung cancer. Anticancer Res. 2010 Jul;30(7):3039-44. PMID 20683052
- [Background] Nishio M, Horai T, Horiike A, Nokihara H, Yamamoto N, Takahashi T, Murakami H, Yamamoto N, Koizumi F, Nishio K, Yusa W, Koyama N, Tamura T. Phase 1 study of lenvatinib combined with carboplatin and paclitaxel in patients with non-small-cell lung cancer. Br J Cancer. 2013 Aug 6;109(3):538-44. doi: 10.1038/bjc.2013.374. Epub 2013 Jul 16. PMID 23860537